CLINICAL TRIAL: NCT03579082
Title: A Clinical Trial of Decitabine in Relapse and Refractory Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, The director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx20171211
Record Dates: First submitted 2017-12-14; First posted 2018-07-06 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Decitabine; ORR; TTP; OS; PFS
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): R±DHAP + decitabine:
  decitabine:10mg/d,ivgtt,d(-5)-(-1);R±DHAP:rituximab,375mg/m2,d0,ivgtt;cytarabine,2g/m2,q12h,d2,ivgtt;cisplatin,100mg/m2,used for 3 days,ivgtt;dexamethasone,40mg,d1-4,ivgtt/po.21 days for one cycle.
  Interventions: Drug: Decitabine
- Arm B (No Intervention): R±DHAP:rituximab,375mg/m2,d0,ivgtt;cytarabine,2g/m2,q12h,d2,ivgtt;cisplatin,100mg/m2,used for 3 days,ivgtt;dexamethasone,40mg,d1-4,ivgtt/po.21 days for one cycle.

INTERVENTIONS:
Drug: Decitabine — Given ivgtt
  Other Names: 5-Aza-2'-deoxycytidine
  Arms: Arm A

SUMMARY:
To explore the safety, tolerability and clinical effects of decitabine combined with R±DHAP for patients with replase and refractory Diffuse Large B cell lymphoma.

DETAILED DESCRIPTION:
This is a randomized,controlled,prospective,open,multi-center clinical trial,amied to evaluate the safety, tolerability,and efficacy of decitabine combined with R±DHAP in replase and refractory Diffuse Large B cell lymphoma.A total of 60 patients are planned to be enrolled into the study.Patients with diagnosis of replase and refractory Diffuse Large B cell lymphoma will be into two groups,and be treated with decitabine pluse R±DHAP or only R±DHAP,respectively.The primary end points are objective responder rate(ORR) and time to progression(TTP) and the secondary end points include overall survival(OS) and progression free survival(PFS).

ELIGIBILITY:
Inclusion Criteria:

* age:14-65 years;ECOG rate≤2;expected survival≥3 months
* patients with Diffuse Large B cell lymphoma diagnoesd by histopathology detection;
* patients ever received RCHOP or CHOP chemotherapy but did not receive DHAP
* patients never received radiotherapy
* patients with no chemotherapy contraindications:hemoglobin ≥ 90g/L,absoluate neutrophil count ≥1.5x109/L,blood platelet ≥100x109/L,ALT and AST ≤ 2-fold upper normal limit,serum bilirubin ≤1.5-fold upper normal limit,serum creatinine ≤1.5-fold upper normal limit,serum albumin ≥ 30g/L,normal serofibrinogen;
* at least one measurable nidus;
* no other severe diseases conflict with this project,cardiopulmonary function is basically normal
* the urine or blood pregnancy test of women in childbearing age must be negative in 7 days before follow-up visit;
* applicable for follow-up visit;
* no other antitumor adjoint therapy(including antitumor Chinese medicine,immunotherapy and biotherapy),but double phosphate anti-bone transfer therapy and other symptomatic treatment are acceptable;
* understanding this study and assigning informed consent.

Exclusion Criteria:

* rejecting providing blood preparation;
* allergic to drug in this study and with metabolic block;
* rejecting adopting reliable contraceptive method in pregnancy or lactation period;
* uncontrolled internal medicine disease(including uncontrolled diabetes,severe incompetence cardiac,lung,liver and pancreas）；
* with severe infection;
* with primary or secondary central nervous system tumor invasion;
* with immunotherapy or radiotherapy contraindication;
* ever suffered with malignant tumor;
* having peripheral nervous system disorder or dysphrenia;
* with no legal capacity,medical or ethical reasons affecting research proceeding;
* participating other clinical trials simultaneously;
* adopting other anti-tumor medicine excluding this research;
* the researchers considering it inappropriate to participate in the study.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 months
  Objective Responder Rate
TTP | up to 2 months
  Time TO Progression

SECONDARY OUTCOMES:
OS | up to 2 months
  Overall Survival
PFS | up to 2 months
  Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Zhang, Principal Investigator — The first affilliated hospital of zhengzhou university
Locations (1):
- Oncology Department of The First Affilliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Hu J, Wang X, Chen F, Ding M, Dong M, Yang W, Yin M, Wu J, Zhang L, Fu X, Sun Z, Li L, Wang X, Li X, Guo S, Zhang D, Lu X, Leng Q, Zhang M, Zhu L, Zhang X, Chen Q. Combination of Decitabine and a Modified Regimen of Cisplatin, Cytarabine and Dexamethasone: A Potential Salvage Regimen for Relapsed or Refractory Diffuse Large B-Cell Lymphoma After Second-Line Treatment Failure. Front Oncol. 2021 Jun 18;11:687374. doi: 10.3389/fonc.2021.687374. eCollection 2021. PMID 34222013